CLINICAL TRIAL: NCT03769948
Title: Validating a Clinical Decision Support Algorithm Developed With Demographic, Co-morbidity, and Lab Data to Diagnose, Stage, Prevent, and Monitor a Patient's Diabetic Retinopathy
Brief Title: Clinical Decision Support Algorithm to Predict Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Oklahoma State University Center for Health Sciences (Other)
Collaborators: Oklahoma State University (Other); University of Oklahoma (Other)
Responsible Party: Principal Investigator, William Paiva, Executive Director, Oklahoma State University
Other Study IDs: HR-18-087
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: risk factors for diabetic retinopathy — Demographic variables: gender, race, marital status, urban rural status. Co-morbidity variable: neuropathy, nephropathy, peripheral circulatory, ketoacidosis, hyperosmolarity Lab tests variables: alanine aminotransferase (ALT), albumin serum, anion gap, aspartate aminotransferase, blood urea nitrogen, calcium serum, chloride serum, creatinine serum, glucose serum plasma, hematocrit, hemoglobin, mean corpuscular hemoglobin concentration (MCHC), mean platelet volume (MPV), potassium serum, protein total serum, red blood cell (RBC) count, sodium serum, white blood cell (WBC) count

SUMMARY:
Diabetic retinopathy (DR), a complication of diabetes, is a leading cause of blindness among working-aged adults globally. In its early stages, DR is symptomless, and can only be detected by an annual eye exam. Once the disease has progressed to the point where vision loss has occurred, the damage is irreversible. Consequently, early detection is quintessential in treating DR. Two barriers to early detection are poor patient compliance with the annual exam and lack of access to specialists in rural areas. This research is focused on developing and validating new, cost-effective predictive technologies that can improve early screening of DR. Our overall objective is to develop and implement an entire suite of tools to detect diabetes complications in order to augment care for underserved rural populations in the US and internationally.

ELIGIBILITY:
Inclusion Criteria:

For diabetic patients with DR:

* With 250.xx diabetes and 362.0x DR ICD-9 codes
* All variables are complete within the observation window

For diabetic patients without DR:

* With 250.xx diabetes ICD-9 codes
* Without 362.0x DR ICD-9 codes
* All variables are complete within the observation window

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The cohort will be selected from diabetic patients that have Electronic Medical Records in Harold Hamm Diabetes Center.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Diabetic retinopathy indicator (yes/no) | March, 2019
  Diabetic patients with 362.0x ICD-9 codes are classified as DR patient